CLINICAL TRIAL: NCT03307122
Title: Infant Formula GI Tolerance Evaluation
Brief Title: Gastrointestinal Tolerance Evaluation of an Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17.01.US.INF
Record Dates: First submitted 2017-09-19; First posted 2017-10-11 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Healthy, Full-term Infants Who Are Formula-fed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Infant Formula 1 (Active Comparator): Routine infant formula with probiotic
  Interventions: Other: Routine Infant Formula 1
- Routine Infant Formula 2 (Active Comparator): Routine infant formula with probiotic and prebiotic
  Interventions: Other: Routine Infant Formula 2

INTERVENTIONS:
Other: Routine Infant Formula 1 — Routine infant formula with probiotic
  Arms: Routine Infant Formula 1
Other: Routine Infant Formula 2 — Routine infant formula with probiotic and prebiotic
  Arms: Routine Infant Formula 2

SUMMARY:
Prospective, double-blind, randomized study of 2 infant formulas.

DETAILED DESCRIPTION:
Exclusively formula-fed infants will participate in a 6-week feeding period of an infant formula. Tolerance records will be kept for 2 days at the end of the 6-week period by caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn singleton infant
* Full-term (> 37 weeks gestation)
* Birth weight ≥ 2500 grams and ≤ 4500 grams
* 9-19 days of age on enrollment
* Infant's mother has elected not to breastfeed prior to enrollment and infant has exclusively formula-fed for at least 3days prior to enrollment
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Known or suspected cow-milk allergy
* Currently receiving a specialty infant formula (e.g. extensively hydrolyzed, amino acid-based, metabolic), or soy-based or lactose free infant formula
* Currently not tolerating (as perceived by the caregiver) their formula
* Currently being treated for reflux
* Currently experiencing gastrointestinal or respiratory symptoms secondary to an on-going infection or virus (e.g. gastrointestinal infection, upper respiratory infection, flu)
* Congenital illness or malformation that may affect infant feeding and/or growth
* Any readmission to hospital (except for hyperbilirubinemia) prior to enrollment
* Receiving prescription medication (with exception of treatment for thrush or topical medications) or home remedies, herbal preparations, or rehydration fluids that might affect GI tolerance (vitamin and mineral supplements excepted).
* Infant's family who in the Investigator's assessment cannot be expected to comply with treatment (feeding regimen).
* Participation in another study that has not been approved as a concomitant study by Nestlé Nutrition.

Ages: 9 Days to 19 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Infant GI Symptom Burden | 6 weeks
  Study personnel will administer questionnaire

SECONDARY OUTCOMES:
Stool pattern | 6 weeks
  Caregivers will document on diary records
Spit-up and/or vomiting pattern | 6 weeks
  Caregivers will document on diary records
Crying and fussing duration | 6 weeks
  Caregivers will document on diary records
Formula intake | 6 weeks
  Caregivers will document on diary records
Formula satisfaction questionnaire | 6 weeks
  Study personnel will administer questionnaire
Weight (measured in grams) | Enrollment and 6 weeks
  Study personnel will measure
Length (measured in centimeters) | Enrollment and 6 weeks
  Study personnel will measure
Adverse events | 2 weeks and 6 weeks
  Assessed throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Carvalho, MD, Study Director — Nestle Nutrition
Locations (8):
- United States (8):
  - Avanza Medical Research Center, Pensacola, Florida
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - PediaResearch, Owensboro, Kentucky
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Midsouth Center for Clinical Research, LLC, Memphis, Tennessee
  - Southwest Children's Research Associates, San Antonio, Texas
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: No